CLINICAL TRIAL: NCT05251519
Title: The Efficacy of Derotation Taping on Balance, Performance, Gait, Spasticity and Quality of Life in Femoral Internal Rotation Deformity in Children With Cerebral Palsy
Brief Title: The Efficacy of Derotation Banding on Outcome Measures in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPKT1
Record Dates: First submitted 2022-01-31; First posted 2022-02-22 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Kinesio taping; Cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping Group (KTG) (Experimental): Conventional rehabilitation application will be performed in addition to Kinesio Tex tape derotation taping.
  Interventions: Other: Kinesio Taping
- Conventional Rehabilitation Group (CRG) (Active Comparator): A conventional rehabilitation program will be applied to the patients through a pediatric physiotherapist.
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Kinesio Taping — Derotation taping with Kinesio Tex is applied to the patients through a pediatric physiotherapist.
  Arms: Kinesio Taping Group (KTG)
Other: Conventional Rehabilitation — Conventional rehabilitation program is applied to the patients through a pediatric physiotherapist
  Arms: Conventional Rehabilitation Group (CRG)

SUMMARY:
The aim of the study is to compare the conventional rehabilitation program and derotation taping applied with Kinesio Tex tape in addition to conventional rehabilitation in children with hemiplegic or monoplegic cerebral palsy with femoral internal rotation deformity.

DETAILED DESCRIPTION:
Conventional rehabilitation (CR) practices will be applied to the control group. Conventional rehabilitation (KT) application will be applied to the study group in addition to Kinesio Tex tape derotation banding. With the kinesio tape application, it is aimed to provide economical, ergonomic and effective support to the patients in non-clinical times. It is aimed to evaluate the patients' balance, quality of life, performance test, spasticity level and gait quality.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy aged 4-12 years with unilateral involvement who are hemiplegic or monoplegic
* Cases with Gross Motor Function Classification (GMFCS) level 1 or 2
* Understanding simple commands and signing the consent form

Exclusion Criteria:

* Presence of a static cause of femoral internal rotation deformity
* Situations that may prevent assessments or communication
* Lack of cooperation during work
* Presence of surgery that may affect assessments, such as joint freezing
* Presence of botulinum toxin administration in the last 6 months
* Development of an allergic reaction on the skin to the tape

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
6MWT | Change from Baseline 6MWT at 3 days
  The 6-meter course was mapped as 10 meters in length with a 2-meter acceleration interval and a 6-meter testing interval. There is no scoring range for the 6MWT.
PBBT | Change from Baseline PBBT at 3 days
  PBBT is a 14-item, criterion-referenced measure and examines functional balance in the context of everyday tasks. PBBT is scored between 0 to 56. Higher scores indicate better function.
MAS | Change from Baseline MAS at 3 days
  The Modified Ashworth Scale is a 6-point rating scale for gauging muscle resistance to passive movement. MAS is scored from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity.
EVGS | Change from Baseline EVGS at 3 days
  EVGS was developed to evaluate gait in children with CP using video recordings. It includes 17 variables, and each of these variables can be scored as 0, 1, or 2 based on movement deviation from normal. enced measure and examines functional balance in the context of everyday tasks. EVGS is scored between 0 to 34. Higher scores indicate worse gait function.
KINDL | Change from Baseline KINDL at 3 days
  The KINDL was derived from a conceptual model, in which the four main components of quality of life, namely psychological well-being, social relationships, physical function and everyday life activities, were included in interviews with children. KINDL is scored between 0 to 100. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet İmerci, PhD, Principal Investigator — Muğla Sıtkı Koçman University; İsmet Tümtürk, BSc, Principal Investigator — Ege University
Locations (1):
- Fethiye Private Son Atılım Special Education and Rehabilitation Center, Muğla, Fethiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No